CLINICAL TRIAL: NCT02538900
Title: Low InTensity Exercise Intervention in PAD
Acronym: LITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary McDermott, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00105855; 1R01HL122846-01 (NIH)
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral arterial disease, peripheral artery disease, PAD, exercise
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Individuals collecting the outcome assessment will not be aware of group assignment.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Low-intensity, self-paced walking exercise. Home based exercise.
  Interventions: Behavioral: Exercise
- Group 2 (Experimental): Standard high intensity, ischemic pain-inducing walking exercise. Home based exercise.
  Interventions: Behavioral: Exercise
- Group 3 (Active Comparator): Non-exercising attention control group. Contact with staff at same frequency as exercise groups, but staff deliver information on health not related to exercise.
  Interventions: Other: Attention control

INTERVENTIONS:
Behavioral: Exercise — Participants in one of the exercise intervention groups will attend once weekly sessions at the medical center for the first four weeks of the study (Weeks 1-4, Phase I). During weeks 5-52 (Phase II), they will receive weekly telephone calls from a study coach.
  Arms: Group 1; Group 2
Other: Attention control — Our attention control group controls for the possibility that regular contact with the study team may improve outcomes in participants randomized to the intervention. Participants randomized to the control group will attend weekly one-hour educational sessions at Northwestern University for the first four weeks of the intervention (Phase I). These sessions are on topics of interest to the typical PAD patient and are led by physicians and other health care workers. Topics include Medicare Part D, nutritional supplements, and cancer screening. During Phase II (weeks 5-52), the attention control group will receive weekly telephone calls, lasting 5-15 minutes, with information on a health-related topic.
  Arms: Group 3

SUMMARY:
This proposed study will determine whether a home-based exercise intervention that avoids continuous supervision and exercise-related ischemic pain improves walking performance at 52-week follow-up in people with PAD, compared to an attention control group and compared to a high intensity exercise intervention. In our secondary aims, we will determine whether high intensity exercise improves six-minute walk distance as compared to the attention control group. In secondary aims, we will also determine whether low intensity exercise and high intensity home-based exercise, respectively, improve patient reported outcomes, physical activity, and treadmill walking performance compared to attention control. Our intervention directly addresses two aspects of current practice guidelines that are major barriers to exercise for patients with PAD: 1) the recommendation for supervised exercise and 2) the recommendation for high intensity ischemic-pain inducing walking exercise.

DETAILED DESCRIPTION:
We will randomize 305 PAD participants to one of three parallel arms: Group 1: Low-intensity, self-paced walking exercise; Group 2: Standard high intensity, ischemic pain-inducing walking exercise; Group 3: Non-exercising attention control group. The low and high intensity exercise groups will attend center-based exercise sessions once per week for four weeks followed by transition to an entirely home-based exercise program for an additional 48 weeks (52 weeks total). Coaches will contact participants weekly by telephone after the first four weeks of the intervention. The low and high intensity exercise interventions will use identical self-regulatory and support strategies. However, the low intensity exercise group will be instructed to exercise with minimal to no ischemic leg discomfort and the high intensity group will be instructed to exercise to maximal ischemic leg pain. These two distinct exercise prescriptions will be reinforced during 48 weeks of home-based exercise, using a well-validated behavioral coaching model that can be delivered by telephone once weekly. Our primary outcome is change in six-minute walk distance at 52-week follow-up. If our hypotheses are correct, millions of people with PAD will benefit from this alternative exercise regimen which will be accessible to most of the 8 million people in the U.S. who suffer from PAD.

ELIGIBILITY:
Inclusion Criteria:

All participants will have PAD. PAD will be defined as follows. First, an ABI < or = 0.90 at the baseline study visit is a well-accepted standard for the diagnosis of PAD and will be an inclusion criterion. Second, people with an ABI of >0.90 and < or = 1.00 who experience a 20% ankle systolic pressure drop after the heel-rise test will also be included. Third, potential participants with an ABI > 0.90 who have vascular lab evidence of PAD or angiographic evidence of PAD who have ischemic symptoms during the six-minute walk and/or treadmill exercise stress test will be eligible. In addition to meeting a criterion for PAD, all participants must be symptomatic, defined by one of the following criteria:; a) ischemic leg symptoms (primarily assessed with the San Diego Claudication Questionnaire); b) report ischemic leg symptoms at the end of the six-minute walk; c) report ischemic leg symptoms at the end of the baseline treadmill stress test; d) walking impairment questionnaire results, e) interview with the potential participant about the presence and nature of leg symptoms during walking activity.

Exclusion Criteria:

1. Above or below knee amputation, critical limb ischemia, wheelchair confinement, or foot ulcer.
2. Individuals whose walking is limited by a condition other than PAD.
3. > Class II NYHA heart failure or angina. Increase in angina, angina at rest, or abnormal baseline treadmill stress test.
4. Major surgery including lower extremity revascularization or orthopedic surgery during the prior three months or anticipated in the next twelve months.
5. Major medical illness including renal disease requiring dialysis, lung disease requiring oxygen other than at night, or cancer (other than non-melanoma skin cancer) requiring treatment in the prior three years. Potential participants may still qualify if they have had treatment for early stage cancer in the previous three years and the prognosis is excellent.
6. Mini-mental status examination score <23, dementia, or psychiatric illness including severe depression or anxiety. Investigator discretion may be used to allow some people with an MMSE below 23 to participate if the investigator determines there is another reason for their lower score, including lack of sufficient familiarity with the English language or lack of sufficient education to achieve a score of 23 or higher.
7. Currently walking regularly for exercise at a level comparable to the amount of exercise prescribed in the intervention.
8. Current or recent (within 3 months) participation in another clinical trial or cardiac rehabilitation. For a clinical trial of a stem cell or gene therapy intervention, potential participants will be potentially eligible immediately after the final study visit for the clinical trial, so long as long as at least six months has passed since the participant received their final treatment in the stem cell or gene therapy intervention. For a clinical trial involving open-label therapy in which the treatment is not related to functional performance and will not change during the LITE Trial, participants may still qualify for the LITE Trial based on investigator discretion.
9. Individuals with PAD who have a history of lower extremity revascularization and have a normal ABI.
10. Individuals who are not able to walk for exercise at a sufficiently slow pace to avoid ischemic leg symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2015-06; Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott, MD, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Ochsner Baptist, Tulane University, New Orleans, Louisiana
  - University of Minnesota, Minneapolis, Minnesota
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Whipple MO, Xu S, Zhang D, Guralnik JM, Spring B, Tian L, Treat-Jacobson D, Zhao L, Criqui MH, McDermott MM. Home-Based Exercise and Patient-Reported Outcome Measures in Peripheral Artery Disease: The LITE Randomized Clinical Trial. Am J Cardiol. 2025 Jun 1;244:41-47. doi: 10.1016/j.amjcard.2025.02.027. Epub 2025 Feb 26. PMID 40020770
- [Derived] Hammond MM, Spring B, Rejeski WJ, Sufit R, Criqui MH, Tian L, Zhao L, Xu S, Kibbe MR, Leeuwenburgh C, Manini T, Forman DE, Treat-Jacobson D, Polonsky TS, Bazzano L, Ferrucci L, Guralnik J, Lloyd-Jones DM, McDermott MM. Effects of Walking Exercise at a Pace With Versus Without Ischemic Leg Symptoms on Functional Performance Measures in People With Lower Extremity Peripheral Artery Disease: The LITE Randomized Clinical Trial. J Am Heart Assoc. 2022 Aug 2;11(15):e025063. doi: 10.1161/JAHA.121.025063. Epub 2022 Jul 27. PMID 35894088
- [Derived] Slysz JT, Rejeski WJ, Treat-Jacobson D, Bazzano LA, Forman DE, Manini TM, Criqui MH, Tian L, Zhao L, Zhang D, Guralnik JM, Ferrucci L, Kibbe MR, Polonsky TS, Spring B, Sufit R, Leeuwenburgh C, McDermott MM. Sustained physical activity in peripheral artery disease: Associations with disease severity, functional performance, health-related quality of life, and subsequent serious adverse events in the LITE randomized clinical trial. Vasc Med. 2021 Oct;26(5):497-506. doi: 10.1177/1358863X21989430. Epub 2021 Apr 8. PMID 33829920
- [Derived] McDermott MM, Spring B, Tian L, Treat-Jacobson D, Ferrucci L, Lloyd-Jones D, Zhao L, Polonsky T, Kibbe MR, Bazzano L, Guralnik JM, Forman DE, Rego A, Zhang D, Domanchuk K, Leeuwenburgh C, Sufit R, Smith B, Manini T, Criqui MH, Rejeski WJ. Effect of Low-Intensity vs High-Intensity Home-Based Walking Exercise on Walk Distance in Patients With Peripheral Artery Disease: The LITE Randomized Clinical Trial. JAMA. 2021 Apr 6;325(13):1266-1276. doi: 10.1001/jama.2021.2536. PMID 33821898

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 116 | 124 | 65
Completed | 96 | 106 | 48
Not Completed | 20 | 18 | 17
Not completed — Death | 2 | 2 | 2
Not completed — Withdrawal by Subject | 18 | 16 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 116 | 124 | 65 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (10.1) | 68.8 (8.7) | 69.5 (10.1) | 69.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 60 | 32 | 146
  Male | 62 | 64 | 33 | 159
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 0 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 65 | 81 | 35 | 181
  White | 45 | 41 | 28 | 114
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 116 | 124 | 65 | 305
Ankle-brachial index [Mean (Standard Deviation); unit: ratio] | 0.66 (0.17) | 0.67 (0.15) | 0.67 (0.15) | 0.66 (0.16)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (6.7) | 31.1 (7.3) | 30.8 (7.3) | 30.7 (7.1)
Six-min walk distance [Mean (Standard Deviation); unit: meters] | 326 (99) | 329 (101) | 328 (87) | 328 (97)

OUTCOME MEASURES:

1. Primary Outcome: Six-minute Walk Distance
Description: In the six-minute walk, participants walk back and forth along a 100-ft hallway for six minutes after standardized instructions to complete as many laps as possible. Distance covered in six minutes is recorded.
Time Frame: change from baseline to week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 116 | 124 | 65
meters | -6.4 [-21.5 to 8.8] | 34.5 [20.1 to 48.9] | -15.1 [-35.8 to 5.7]

2. Secondary Outcome: Six-minute Walk Distance
Description: as for outcome 1
Time Frame: change from baseline to week 26
Reporting Status: Not Posted

3. Secondary Outcome: Maximal Treadmill Walking Time
Description: In the treadmill walking test, participants walk on either a gardner or modified gardner protocol until they stop the test. Time walked is recorded
Time Frame: change from baseline to week 52
Reporting Status: Not Posted

4. Secondary Outcome: Physical Activity Levels
Description: ActiGraph measured physical activity
Time Frame: Change from baseline to week 52
Reporting Status: Not Posted

5. Secondary Outcome: Walking Impairment Questionnaire (WIQ) Distance and Speed Score.
Description: The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed.
Time Frame: change from baseline to week 52
Reporting Status: Not Posted

6. Secondary Outcome: Health-related Quality of Life Measure
Description: The SF-36 physical functioning score will be used to measure quality of life.
Time Frame: change from baseline to week 52
Reporting Status: Not Posted

7. Secondary Outcome: Adherence to Intervention
Description: Adherence is defined as the proportion achieving at least 80% of the prescribed exercise frequency and duration during the final month of the intervention.
Time Frame: from baseline to week 52
Reporting Status: Not Posted

8. Secondary Outcome: Change in Muscle Biopsy Measures of Mitochondrial Oxidative Metabolism and Oxidative Stress.
Description: Muscle tissue will be collected at baseline and follow up to measures Change in muscle biopsy measures of mitochondrial oxidative metabolism and oxidative stress.
Time Frame: change from baseline to week 52
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Qualitative Assessment
Description: We will use qualitative methods to explore participants' perceptions of the exercise interventions in the high and low-intensity exercise groups, respectively.
Time Frame: At 52 week follow up
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Physical Activity Levels Over Seven Days
Description: ActiGraph
Time Frame: 26 week follow-up.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: WIQ Distance and Speed Score
Description: The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed.
Time Frame: 26 week follow-up
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Health Related Quality of Life
Description: SF-36 physical functioning score.
Time Frame: 26 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Adherence to Assigned Intervention
Description: as for outcome 7
Time Frame: 26 weeks.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected monthly through out the 12-month intervention period.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 2/116 | 2/124 | 2/65
Serious Adverse Events (participants affected / at risk) | 43/116 | 40/124 | 19/65
Other Adverse Events (participants affected / at risk) | 34/116 | 42/124 | 29/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=116) | Group 2 (N=124) | Group 3 (N=65)
Lower extremity revascularization (Cardiac disorders) | 8 (8) | 9 (9) | 2 (2)
Infection (Infections and infestations) | 6 (6) | 11 (11) | 1 (1)
Chest pain (General disorders) | 5 (5) | 4 (4) | 5 (5)
Ischemic heart disease (Cardiac disorders) | 4 (4) | 4 (4) | 0 (0)
Abdominal problem (General disorders) | 3 (3) | 5 (5) | 0 (0)
Diabetes (General disorders) | 3 (3) | 2 (2) | 2 (2)
GI bleed (General disorders) | 1 (1) | 4 (4) | 2 (2)
Critical limb ischemia (Vascular disorders) | 2 (2) | 4 (4) | 0 (0)
Fall or fracture (General disorders) | 3 (3) | 1 (1) | 2 (2)
Pulmonary event (General disorders) | 5 (5) | 0 (0) | 1 (1)
Stroke or cerebral hemorrhage (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1)
Elective surgery (General disorders) | 3 (3) | 1 (1) | 1 (1)
Syncope (General disorders) | 1 (1) | 2 (2) | 2 (2)
Arrhythmia (General disorders) | 2 (2) | 2 (2) | 0 (0)
Coronary revascularization (General disorders) | 3 (3) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0)
Lightheaded (General disorders) | 2 (2) | 1 (1) | 1 (1)
Venous thromboembolism (General disorders) | 2 (2) | 2 (2) | 0 (0)
Carotid revascularization (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Headache (General disorders) | 3 (3) | 0 (0) | 0 (0)
Hypertension (General disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal infection (General disorders) | 0 (0) | 1 (1) | 0 (0)
Acute renal failure (General disorders) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (General disorders) | 0 (0) | 2 (2) | 0 (0)
Cancer (General disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (General disorders) | 0 (0) | 0 (0) | 2 (2)
Dehydration (General disorders) | 1 (1) | 1 (1) | 0 (0)
Esophageal problem (General disorders) | 1 (1) | 0 (0) | 1 (1)
PAD (General disorders) | 0 (0) | 2 (2) | 0 (0)
Angina (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bowel obstruction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Complication from angiogram (General disorders) | 0 (0) | 1 (1) | 0 (0)
Complication from medical procedure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Congestive heart failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Diagnostic testing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Electrolyte problem (General disorders) | 0 (0) | 1 (1) | 0 (0)
Medication side effect (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status (General disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal (General disorders) | 1 (1) | 0 (0) | 0 (0)
Neurologic problem (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusions (General disorders) | 1 (1) | 0 (0) | 0 (0)
Psychiatric (General disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular problem (General disorders) | 0 (0) | 1 (1) | 1 (1)
Ulcer (General disorders) | 0 (0) | 0 (0) | 1 (1)
Weight loss (General disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=116) | Group 2 (N=124) | Group 3 (N=65)
New or increased chest discomfort during activity or exercise (General disorders) | 9 (11) | 16 (23) | 8 (14)
New or increased shortness of breath during activity or exercise (General disorders) | 13 (21) | 24 (38) | 19 (30)
New or increased dizziness or generalized weakness during activity or exercise (General disorders) | 23 (25) | 21 (28) | 22 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT02538900/Prot_SAP_000.pdf